CLINICAL TRIAL: NCT01239004
Title: A 12-Week, Double-Blind, Randomized, Placebo-Controlled Study to Assess the LDL Cholesterol Lowering and Anti-Hyperglycemic Efficacy of Welchol® (Colesevelam) in Subjects With Impaired Fasting Glucose Who Are Taking Niaspan® (Niacin) for Dyslipidemia
Brief Title: Colesevelam Treatment for Impaired Fasting Glucose During Niacin Therapy
Acronym: CERTAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radiant Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Welchol-Niaspan 001
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Dyslipidemia; Hyperlipidemia; Hyperglycemia
Keywords: dyslipidemia; hyperlipidemia; hyperglycemia; impaired fasting glucose
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias; Hyperglycemia | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Colesevelam (Experimental)
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Placebo — 6 tablets daily, with up to 2000 mg niacin and 325 mg aspirin daily, for 12 weeks
  Arms: Placebo
Drug: Colesevelam — 6 tablets (3750 mg total) daily, with up to 2000 mg niacin and 325 mg aspirin daily, for 12 weeks
  Other Names: Welchol
  Arms: Colesevelam

SUMMARY:
The present study will assess the low-density lipoprotein cholesterol (LDL-C) lowering effect of colesevelam as an adjunct to niacin for the improvement of lipids and glycemic control in dyslipidemic subjects with impaired fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Non-HDL-C ≥100 mg/dL and ≤220 mg/dL at Visits 1 and 2.
3. FPG ≥90 mg/dL and ≤145 mg/dL, at Visits 1 and 2.
4. HDL-C <60 mg/dL at Visits 1 and 2, regardless of gender.
5. Untreated dyslipidemia, or statin treatment only with equipotency to atorvastatin ≤40 mg daily for at least 12 weeks prior to Screening Visit 1 and without change or initiation prior to randomization

Exclusion Criteria:

1. Known intolerance to niacin or bile acid-sequestering drugs or aspirin.
2. Any contraindication to a study medication (niacin, aspirin or colesevelam).
3. History of dysphagia, swallowing disorders or intestinal motility disorders.
4. History of pancreatitis.
5. Fasting TG >500 mg/dL at Visits 1 and 2
6. Currently taking medication for diabetes mellitus, Type 1 or 2,or currently taking glucose-lowering drugs (e.g. metformin) for any other indication.
7. Currently taking drugs that may affect glycemic and/or lipid control (e.g., beta-blockers, etc.) if started within the 12 weeks prior to Visit 1, or prior to randomization. This does not apply to dietary supplements.).
8. Body mass index (BMI) >40 kg/m2.
9. History of acute myocardial infarction, unstable angina, transient ischemic attacks, stroke or revascularization procedure within the 3 months prior to Visit 1 or prior to randomization.
10. Use of prescription strength niacin, bile acid sequestrants, fibrates or omega-3 fatty acids within 8 weeks prior to Visit 1 or prior to randomization. This does not apply to dietary supplements.
11. Unwilling to abstain, during the study, from weight-loss drugs (including over-the-counter) or weight-loss programs during the study.
12. Current use, or intended use during the study, of cyclic hormones (e.g., oral or vaginal contraceptives and estrogen replacement therapy).
13. Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential not using an acceptable method of contraception. Acceptable methods include intrauterine device, cervical diaphragm plus spermicide, female condom plus spermicide, or partner's use of condoms plus spermicide. Partner's vasectomy only or use of condoms or spermicide only are not considered acceptable forms of birth control.
14. Current use, or intended use during the study of cyclosporine.
15. Recent history (past 12 months) of illicit drug use or excessive ethanol use. Excessive ethanol use will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
16. Exposure to any investigational agent within 30 days prior to Visit 1, and prior to randomization.
17. Individual has a condition the Investigator believes would interfere with his ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol (LDL-C) | 12 weeks
  The primary efficacy endpoint will be the mean percent change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in LDL-C. It will be measured as part of the fasting lipid panel at Visits 1, 2, 3, 7, and 8/ET (Weeks -6 to -2, -1, 1, 10 and 12/ET).

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG) | 12 weeks
  The principal secondary efficacy endpoint is the mean change in FPG from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12).
NMR Lipid subfractions and lipoprotein-IR score | 12 weeks
  A secondary efficacy endpoint is the mean change from baseline (Week 1) to end-of-treatment(Week 12) in NMR Lipid subfractions and lipoprotein-IR score.
Hemoglobin A1C (HbA1C) | 12 weeks
  A secondary efficacy endpoint is the mean change from baseline (Week 1) to end-of-treatment(Week 12) in HbA1c.
Fructosamine | 12 weeks
  A secondary efficacy endpoint is the mean change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in fructosamine.
High sensitivity c-reactive protein (hs-CRP) | 12 weeks
  A secondary efficacy endpoint is the mean change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in hs-CRP.
Niacin-related flushing | 12 weeks
  Niacin-associated flushing will be measured using a visual analog scale (VAS)at Weeks 2,4,6,10 and 12.
Homeostasis model assessment of insulin resistance (HOMA-IR) score | 12 weeks
  A secondary efficacy endpoint is the mean change from baseline (Week 1) to end-of-treatment (Week 12) in HOMA-IR.
High-density lipoprotein cholesterol (HDL-C) | 12 weeks
  A secondary endpoint is the mean percent change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in HDL-C.
Non-high-density lipoprotein cholesterol (non-HDL-C) | 12 weeks
  A secondary endpoint is the mean percent change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in non-HDL-C.
Total Cholesterol (TC) | 12 weeks
  A secondary endpoint is the mean percent change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in TC.
Triglycerides (TG) | 12 weeks
  A secondary endpoint is the mean percent change from baseline (average of Weeks -1 and 1) to end-of-treatment (average of Weeks 10 and 12) in TG.
Fasting Insulin | 12 weeks
  A secondary efficacy endpoint is the mean change from baseline (Week 1) to end-of-treatment (Week 12) in fasting insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD, FACC, Principal Investigator — Executive Medical Director, Radiant Research
Locations (4):
- United States (4):
  - Radiant Research, Chicago, Illinois
  - Kansas City, Kansas
  - Minneapolis, Minnesota
  - St Louis, Missouri